CLINICAL TRIAL: NCT02329405
Title: PXR-aktivaation Vaikutus Maksan Rasvoittumiseen
Brief Title: The Effects of PXR Activation on Hepatic Fat Content
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Rifa-Stea; 2014-003422-41 (EudraCT Number)
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifampicin (Experimental): Rifampicin 600 mg tablet once a day orally for a week.
  Interventions: Drug: Rifampicin
- Placebo (Placebo Comparator): Placebo tablet once a day orally for a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifampicin
  Other Names: Rifampin
  Arms: Rifampicin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study investigates the effects of pregnane X receptor (PXR) activation on hepatic fat content in healthy volunteers. Rifampicin (an antibiotic and also an efficient PXR activator) and placebo will be given for a week to volunteers. Hepatic fat content is measured with magnetic resonance imaging and blood samples are collected at the end of each study arm. The investigators' hypothesis is that rifampicin causes accumulation of fat to the liver.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Body mass index (BMI) 18.5-25 kg/m2

Exclusion Criteria:

* Systolic blood pressure over 150 mmHg
* Any continuous medication (hormonal intrauterine device is permitted)
* Any significant medical condition
* Insensitivity to rifampicin
* Pregnancy and lactation
* Previous difficult venipuncture
* Alcohol and medicine abuse and drug use
* Participation to any other pharmaceutical trial within on month of screening
* Claustrophobia
* Metal and other implants which are contraindications to MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Hepatic fat fraction | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Rahunen R, Kummu O, Koivukangas V, Hautajarvi H, Hakkola J, Rysa J, Hukkanen J. Pregnane X Receptor-4beta-Hydroxycholesterol Axis in the Regulation of Overweight- and Obesity-Induced Hypertension. J Am Heart Assoc. 2022 Mar 15;11(6):e023492. doi: 10.1161/JAHA.121.023492. Epub 2022 Mar 1. PMID 35229613